CLINICAL TRIAL: NCT03868007
Title: Protective Effects of Remote Ischemic Conditioning in Elderly With Acute Ischemic Stroke Complicating Acute Coronary Syndrome: A Single-center Randomised Controlled Trial
Brief Title: Protective Effects of RIC in Elderly With Acute Ischemic Stroke Complicating Acute Coronary Syndrome
Acronym: RIC-ACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RIC-ACS
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Elderly Patients; Acute Ischemic Stroke; Acute Coronary Syndrome
Keywords: remote ischemic conditioning; elderly; acute ischemic stroke; Acute Coronary Syndrome
MeSH Terms: conditions — Ischemic Stroke; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The RIC and sham procedure were performed by using identical devices with different cuff pressures (200mmHg versus 60 mmHg). Patients, investigators, and raters were all blinded to the treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): Patients with AIS complicating ACS who were eligible for this study received standardized medical treatment and secondary prevention, including antiplatelets, low molecular weight heparin for anticoagulation，statins for lipid-lowering and stabilizing plaque, nitrates for vascular expansion and cardiocerebrovascular risk factors management. Administration of antihypertensive, antidiabetic or other agents were elective at the discretion of the treating physician according to the conditions of the patients. In addition, patients underwent RIC twice daily for 14 days.And the RIC procedure during which bilateral arm cuffs are inflated to a pressure of 200mmHg for five cycles of 5 min followed by 5 min of relaxation of the cuffs.
  Interventions: Device: RIC
- sham-RIC group (Sham Comparator): Patients with AIS complicating ACS who were eligible for this study received standardized medical treatment and secondary prevention, including antiplatelets, low molecular weight heparin for anticoagulation，statins for lipid-lowering and stabilizing plaque, nitrates for vascular expansion and cardiocerebrovascular risk factors management. Administration of antihypertensive, antidiabetic or other agents were elective at the discretion of the treating physician according to the conditions of the patients. In addition, patients underwent sham-RIC twice daily for 14 days.And the sham-RIC procedure during which bilateral arm cuffs are inflated to a pressure of 60mmHg for five cycles of 5 min followed by 5 min of relaxation of the cuffs.
  Interventions: Device: sham-RIC

INTERVENTIONS:
Device: RIC — The RIC procedure during which bilateral arm cuffs are inflated to a pressure of 200mmHg for five cycles of 5 min followed by 5 min of relaxation of the cuffs.
  Arms: RIC group
Device: sham-RIC — The sham-RIC procedure during which bilateral arm cuffs are inflated to a pressure of 60mmHg for five cycles of 5 min followed by 5 min of relaxation of the cuffs.
  Arms: sham-RIC group

SUMMARY:
Remote ischemic conditioning (RIC) is a noninvasive strategy in which one or more cycles of brief and transient limb ischemia confers protection against prolonged and severe ischemia in distant organs.This study aimed to investigate whether RIC is safe and effective in patients with AIS complicating ACS

DETAILED DESCRIPTION:
Remote ischemic conditioning (RIC) is a noninvasive strategy in which one or more cycles of brief and transient limb ischemia confers protection against prolonged and severe ischemia in distant organs (e.g., brain and heart).It has been demonstrated to be an effective strategy to reduce plasma myocardial enzyme, infarct volume, and incidence of post-ACS heart failure in patients with ACS. Additionally, recent studies have found that RIC was safe and feasible in patients with AIS even in those caused by large artery occlusion and treated with reperfusion therapy, and it might benefit AIS patients by reducing the risk of brain tissue infarction and improving functional outcomes. To date, however, it is still unknow whether RIC, a systematic protective strategy, could benefit patients with AIS complicating ACS.This study aimed to investigate whether RIC is safe and effective in patients with AIS complicating ACS.

ELIGIBILITY:
Inclusion Criteria:

* age≥60yo
* AIS within 24 hours after symptom onset which meet the diagnostic criteria for acute ischemic stroke of the 2013th ASA guidelines, AIS was defined as a clinical episode of neurological dysfunction caused by focal cerebral infarction that can be detected on imaging(e.g.,computed tomography or magnetic resonance imaging of head)
* ACS within 24 hours of stroke onset , and ACS contains ST-segment elevation myocardial infarction, non-ST-elevation myocardial infarction, unstable angina and it was defined when there is a rise and/or fall of plasma cardiac biomarkers (e.g., myocardial enzyme，cardiac troponin I), along with supportive evidence in the form of typical symptoms (e.g., chest pain), suggestive electrocardiographic changes, or imaging evidence of new loss of viable myocardium or new regional wall motion abnormality
* The patients missed the opportunity of or contradicted to reperfusion therapy (i.e., intravenous thrombolysis and endovascular treatments) for both AIS and ACS.
* Informed consent obtained

Exclusion Criteria:

* Unstable vital signs
* Prior ipsilateral stroke with residual deficits
* AIS caused by cardioembolism, suspicious arterial dissection, intracranial sinus thrombolysis, vasculitis, and moyamoya disease.
* Intracranial bleeding.
* Advanced malignancy.
* Uncontrolled hypertension (defined as systolic blood pressure ≥200 mm Hg despite medications at enrollment).
* Any vascular, soft tissue, or orthopedic injury (eg, superficial wounds and fractures of the arm) that contraindicated bilateral arm ischemic preconditioning.
* Peripheral vascular disease that affecting the upper limbs' arteries
* Any disorder that could potentially increase pre-stroke myocardial enzyme concentrations (eg, percutaneous coronary intervention or myocardial infarction within the previous 6 weeks)
* Coronary artery stenosis requiring coronary bypass surgery for the index event within 3 months; or severe heart failure requiring mechanical ventilation or use of an intra-aortic balloon pump
* Taking drugs in the study period or are participating in other clinical trials.
* Severe psychiatric disease.
* Patients who cannot keep treatment or follow-up.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2022-01-08 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCEs) | from baseline to 3 months after therapy
  MACCEs defined as all cause of death and recurrence of cardiac and cerebrovascular ischemic events within 3 months after randomization

SECONDARY OUTCOMES:
the proportion of patients achieving functional independence | from baseline to 3 months after therapy
  Functional independence is defined as modified Ranks scale [mRS] ≤2 points
the national institutes of health stroke (NIHSS) score | changes from baseline to 7 days, 14 days ,30 days, 90 days after therapy
  National Institute of Health Stroke Scale (NIHSS) is considered as a standardized assessment of neurological functions in the acute phase of stroke, and it is generally used to quantify patient's neurological impairments on 15 items in 11 fields of different neurological status.The score of the scale ranges from 0 to 42.And higher score indicates worse neurological function.The NHISS will be assessed by certified study investigator, who is blinded to the treatment assignment.
plasma hypersensitive C-reactive protein（hs-CRP） level | changes from baseline to 2 weeks after therapy
  Blood samples were drawn from the cubital vein after enrolling into this study and two weeks after randomization. These samples were centrifuged immediately collection, and serum hs-CRP level were examined in fresh plasma samples.
global registry of acute coronary events (GRACE) score | changes from baseline to 7 days, 14 days ,30 days, 90 days after therapy
  For each patient, GRACE score was calculated by using specific variables collected at admission. Patients were classified into 3 categories low (1-108), intermediate (109-140), and high (>140), according to the GRACE score
modified Rankin scale（mRs） | changes from baseline to 7 days, 14 days ,30 days, 90 days after therapy
  this scale is to evaluate the neurological function，it ranges form 0 to 6, the lower score means better neurological outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li S, Xing X, Wang L, Xu J, Ren C, Li Y, Wang J, Liu Z, Zhao H, Zhao W, Ji X. Remote ischemic conditioning reduces adverse events in patients with acute ischemic stroke complicating acute myocardial infarction: a randomized controlled trial. Crit Care. 2024 Jan 2;28(1):5. doi: 10.1186/s13054-023-04786-y. PMID 38167175